CLINICAL TRIAL: NCT07180212
Title: The Guiding Value of Urinary Tumor DNA Testing in Cystoscopy for High-Risk/Very High-Risk Non-Muscle-Invasive Bladder Cancer: An Open-Label, Randomized Controlled, Multicenter Clinical Study (Truce-LB02)
Brief Title: Guiding Value of Urinary Tumor DNA Testing in Cystoscopy for High-Risk/Very High-Risk Non-Muscle-Invasive Bladder Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Truce-LB02
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer; Liquid Biopsy; Cystoscopy
Keywords: bladder cancer; liquid biopsy; cystoscopy; urine tumor DNA
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will undergo urine tumor DNA (utDNA) testing and urine cytology every 3 months, and cystoscopy once per year. If either utDNA or urine cytology is positive, an additional cystoscopy will be performed. If urine cytology is positive but cystoscopy is negative, or if two consecutive utDNA tests are positive while cystoscopy remains negative, participants will undergo computed tomography urography (CTU) to evaluate the upper urinary tract.
  Interventions: Diagnostic Test: utDNA testing + Urine Cytology
- Arm B (Active Comparator): Participants will undergo cystoscopy and urine cytology every 3 months. If urine cytology is positive but cystoscopy is negative, participants will undergo computed tomography urography (CTU) to evaluate the upper urinary tract.
  Interventions: Diagnostic Test: Cystoscopy + Urine Cytology

INTERVENTIONS:
Diagnostic Test: utDNA testing + Urine Cytology — Participants undergo urine tumor DNA (utDNA) testing and urine cytology every 3 months, and cystoscopy once per year. If either utDNA or urine cytology is positive, an additional cystoscopy will be performed. If urine cytology is positive but cystoscopy is negative, or if two consecutive utDNA tests are positive while cystoscopy remains negative, participants will undergo computed tomography urography (CTU) to evaluate the upper urinary tract.
  Arms: Arm A
Diagnostic Test: Cystoscopy + Urine Cytology — Participants undergo cystoscopy and urine cytology every 3 months as per standard high-risk NMIBC surveillance. If urine cytology is positive but cystoscopy is negative, participants will undergo computed tomography urography (CTU) to evaluate the upper urinary tract.
  Arms: Arm B

SUMMARY:
Non-muscle-invasive bladder cancer (NMIBC) is usually treated with surgery to remove the tumor (transurethral resection of bladder tumor, or TURBT), often followed by bladder-instilled medications to reduce the chance of the cancer coming back. Even with this treatment, high-grade NMIBC can return or progress, so patients need regular check-ups, usually with cystoscopy (a camera examination of the bladder) and urine cytology.

Cystoscopy is effective but invasive, can cause discomfort, and carries risks such as infection and bleeding. This makes follow-up costly and sometimes burdensome for patients.

This study is testing whether a urine tumor DNA (utDNA) test - a type of "liquid biopsy" that detects cancer-related DNA changes in urine - can help guide the timing of cystoscopy for people with high-risk or very high-risk NMIBC. utDNA testing is non-invasive and has shown high accuracy in detecting bladder cancer, sometimes spotting signs of recurrence earlier than standard methods.

By combining utDNA testing with cystoscopy, we hope to safely reduce the number of unnecessary cystoscopies without missing cancer recurrences. The study will evaluate whether this approach can make bladder cancer follow-up more comfortable, more precise, and more efficient.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 18 years or older.
2. Histologically confirmed high-risk or very high-risk non-muscle-invasive urothelial carcinoma (NMIBC) of the bladder, as defined by the EAU 2025 NMIBC guidelines, or bladder tumors in which high-risk/very high-risk NMIBC constitutes more than 50% of the pathological composition, diagnosed within the past 2 years, with no evidence of muscle-invasive bladder cancer or metastatic disease.
3. Prior to enrollment, participants must have undergone either:

A.Second transurethral resection of bladder tumor (re-TURBT), or B.Complete initial TURBT with negative basal margins, peripheral margins, and multiple site biopsies, with pathological specimens including detrusor muscle and showing no residual tumor, and negative urine cytology at 2 weeks post-surgery.

Exclusion Criteria:

1.History of upper urinary tract malignancy (ureter or renal pelvis) within the past 5 years or concurrent diagnosis of upper urinary tract urothelial carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 24 months from randomization.
  Time from randomization to the first histologically confirmed intravesical tumor recurrence (any grade/stage).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months from randomization.
  Time from randomization to pathologic progression to muscle-invasive bladder cancer (≥T2), any newly diagnosed upper tract urothelial carcinoma (UTUC), distant metastasis from urothelial carcinoma, radical cystectomy or nephroureterectomy performed for oncologic progression, or urothelial carcinoma-specific death, whichever occurs first.
Diagnostic/Prognostic Performance of utDNA | From randomization to 24 months.
  Predictive value of utDNA for subsequent recurrence/progression, including sensitivity, specificity, PPV, NPV, time-dependent AUC/C-index at 12 and 24 months, and hazard ratios from Cox models adjusted for prespecified covariates.

CONTACTS AND LOCATIONS:
Locations (1):
- The second hospital of Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to patient privacy concerns and institutional restrictions.